CLINICAL TRIAL: NCT07251010
Title: Phrenoesophageal Ligament Reconstruction With Mesh: A New Approach to Hiatal Hernia Repair (Alinasser's Technique) for Adult Patients With Symptomatic Hiatus Hernia: A Randomized Controlled Trial
Brief Title: Phrenoesophageal Ligament Reconstruction With Mesh
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Trial Aseer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHC-RCT-4-2025; AHC-RCT-4-2025 (Other: ClinicalTrialAseer)
Record Dates: First submitted 2025-09-24; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hiatus Hernia; Gastreoesophageal Reflux Disease
Keywords: hiatus hernia; Gastroesophageal reflux disease
MeSH Terms: conditions — Hernia, Hiatal; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic approach (Standard of Care) (Experimental): Standard Surgical Procedure Hiatal hernia repair no Mesh
  Interventions: Procedure: Classic approach
- Hiatal Hernia Repair and Phrenoesophageal Ligament Reconstruction with Mesh (Alinasser technique) (Experimental): A New Approach
  Interventions: Procedure: Phrenoesophageal Ligament Reconstruction with Mesh: A New Approach to Hiatal Hernia Repair (Alinasser's Technique)

INTERVENTIONS:
Procedure: Phrenoesophageal Ligament Reconstruction with Mesh: A New Approach to Hiatal Hernia Repair (Alinasser's Technique) — Alinasser's technique of laparoscopic hiatal hernia repair (LHHR) is carried out, follow same steps of classical approach except before closing the crura A non-absorbable mesh (≈2.0 x 10.0 cm) is sutured to the esophagus( lower mediastinal esophagus) , just above the hiatus by four 2-0 prolene stitches. The continuity of the mesh is then fixed just below the hiatus anteriorly on the abdominal face of diaphragm by four 2-0 prolene stitches. About half of the mesh is fixed to the esophagus and the other half is fixed to the diaphragm. If there is no space for mesh fixation on the diaphragm, the left hepatic triangular ligament will be released.
  Arms: Hiatal Hernia Repair and Phrenoesophageal Ligament Reconstruction with Mesh (Alinasser technique)
Procedure: Classic approach — Classic approach of laparoscopic hiatal hernia repair (LHHR) is performed under general anesthesia with the patient in the French position and pneumoperitoneum established at 15 mmHg CO₂. Port placement follows a standardized foregut approach, with a camera port in the epigastrium and additional working ports placed under direct vision. After retracting the left lobe of the liver, the diaphragmatic hiatus is exposed. The stomach and hernia sac are reduced by dividing short gastric vessels and mobilizing the gastric fundus to free the left crus. Circumferential dissection of the hernia sac continues cranially to gain at least 3-5 cm of intraabdominal esophageal length.The diaphragmatic crura are approximated posterior to the esophagus, aided by a calibration tube. If necessary. A posterior 270° Toupét fundoplication is then constructed with interrupted stitches, anchoring the wrap to the esophagus and crura.
  Arms: Classic approach (Standard of Care)

SUMMARY:
Introduction: The phrenoesophageal ligament (PEL) is a crucial structure that attaches the esophagus to the diaphragm, allowing for independent movement during respiration and swallowing. The ligament provides flexibility and strength, maintaining the integrity of the esophageal hiatus while accommodating pressure changes during breathing and swallowing. It consists of two limbs. The upper limb attaches the esophagus to the superior surface of the diaphragm, extending through the hiatus t'o insert into the esophagus 2-3 cm above it. The Lower Limb attaches the cardiac region of the stomach to the inferior surface of the diaphragm at the cardiac notch of the stomach. Failure and weakness of the PEL can predispose to esophageal HH and GERD symptoms. Understanding its anatomy is essential for the surgical management of hiatal hernia and GERD.

Purpose: To investigate the effectiveness and safety of a new technique for hiatal hernia repair (Alinasser's Technique of LHHR) using a mesh fixed to both the esophagus and crura, mimicking PEL, with a focus on reducing recurrence rates and improving patient outcomes. Methods: A randomized controlled trial study will be followed. The study will include 60 HH patients who will be randomized into either the intervention group (30 patients) who will undergo the new approach, or the classic group (30 patients) who will undergo the classic approach. Patients in the intervention group will undergo cruroplasty using a new technique (mesh applied like PEL). Importance: A new surgical technique is being applied for management of HH to decrease postoperative recurrence

DETAILED DESCRIPTION:
Diagnosis of GERD, esophagitis, and hiatus hernia:

Preoperative diagnosis We will use the GERD-Health-Related Quality of Life (GERD-HRQL) questionnaire to evaluate symptoms of GERD [11]. Preoperative assessment to diagnose HH by upper GIT endoscopy and a barium meal test in reverse Trendelenburg position. The Los Angeles system will be used for grading esophagitis [12]. 24 pH and esophageal manometry will be used to assess the esophageal motility and esophageal PH

Surgical technique:

Under general anaesthesia, Alinasser's Technique of LHHR will be carried out in the Frensh position. The pneumoperitoneum was created with CO2 pressures as high as 15 mmHg.

Procedure Position. The patient is positioned the French position, the surgeon stands in-between the legs and the assistants stand on either side of the patient, Steep reverse Trendelenburg positioning is often required. Port placement. We use a standard ports placement for most foregut procedures performed.

This consists of establishment of pneumo-peritoneum using a Veress needle placed at Palmer's point in the left upper abdomen. An 10-mm optical trocar is inserted in the left subcostal position.

Additional ports are placed under direct vision as follows (Figure 1):

* Camera port (10 mm) in epigastric position (midway between the xiphoid process and the umbilicus.
* Assistant (5 mm) port at the left anterior axillary line below the costal margin.
* Surgeon's left hand port (5 mm) in right upper quadrant at the midclavicular line.

  1. Expose the diaphragmatic hiatus by retracting the left lateral segment of the liver.
  2. Reduce stomach and hiatal hernia sac by mobilizing the gastric fundus. Dissection begins with takedown of short gastric vessels and proceeds toward the diaphragmatic hiatus to fully expose the left diaphragmatic crus.
  3. Complete circumferential dissection of the hiatal hernia sac at the level of diaphragmatic hiatus. It is often easiest to gain entry into the proper plane immediately adjacent to the left crus. The correct plane is bloodless and involves division of loose areolar attachments. The right crus is approached by dividing the pars flaccida and dissected until the left crus is visualized. It is important to preserve the integrity of the crura during this phase of the dissection.
  4. The mediastinal dissection continues in a cranial direction to obtain enough intraabdominal esophageal length (minimum 3-5 cm).
  5. A non-absorbable mesh (≈2.0 x 10.0 cm) is sutured to the esophagus, just above the hiatus by four 2-0 prolene stitches. The continuity of the mesh is then fixed just below the hiatus anteriorly on the diaphragm by four 2-0 prolene stitches. About half of the mesh is fixed to the esophagus and the other half is fixed to the diaphragm.
  6. Re-approximation of the diaphragmatic crura is performed posterior to the esophagus using interrupted 0 non-absorbable sutures. A calibration tube is used to judge the approximation limit.
  7. If there is no space for mesh fixation on the diaphragm, the left hepatic triangular ligament will be released.
  8. Toupét fundoplication fashioned by positioning of the fundus posterior to the esophagus.

     Three Interrupted 2-0 sutures are then used to anchor the stomach to the lower esophagus antero-laterally. Then, the left gastric segment is sutured to the esophagus antero-laterally, leaving a gap of 1.5 to 2 cm from the right gastric segment, completing a 270° wrap.
  9. The wrap is then anchored to the hiatus using interrupted 2-0 non-absorbable sutures.

Typically, four sutures are required to anchor the wrap to both the right and left crura as well as the anterior aspect of the diaphragmatic hiatus. The routine postoperative Care is achieved The Primary Outcome is the recurrence rate of hiatal hernia, as assessed by Endoscopy and imaging studies (e.g., barium meal in Trendelenburg position or endoscopy) at 1-2 years follow-up. Secondary Outcomes are the complication rates (e.g., dysphagia, mesh erosion, infection), Operative time, patient satisfaction and quality of life, hospital stay, readmission rate, Reoperation rate, Symptom improvement (e.g., reflux, chest pain), and coast Postoperative management Every day, vital signs such as heart rate, blood pressure, oxygen saturation, and intravenous fluid levels will be documented. Clear oral fluid will be initiated six hours after surgery. In the absence of any formal complaints, patients will be allowed to be discharged from the hospital. Follow up There are scheduled follow-up appointments at1,3,6,12, and 24 months postoperatively. The follow-up consisted of a clinical evaluation including presence of symptoms of GERD (heartburn, regurgitation, epigastric discomfort) or nonspecific symptoms such as dysphagia or vomiting), upper GIT endoscopy, radiographic barium meal in trendlenberge position and abdominal CT for selected patient. Statistical analysis For categorical variables, we utilized percentages and numbers as descriptive statistics, whereas for continuous variables, we used mean and standard deviations. The statistical analyses were conducted using SPSS 26 (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
* Eligibility criteria have been reformatted as follows:

  #Inclusion Criteria:
* Adult patients (≥18 years)
* Symptomatic hiatus hernia
* Primary hiatus hernia
* Not responding to medical treatment

  #Exclusion Criteria:
* Children (<18 years)
* Recurrent hiatus hernia
* Post-bariatric surgery
* Pregnancy
* Crohn's disease
* Emergency surgery cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The recurrence rate of hiatal hernia by imaging and endoscopy | 12 Months Post- surgery
  Imaging-based diagnosis: Most studies utilize radiological evaluation, such as esophagram (fluoroscopic imaging), CT scans, or barium swallow tests, to detect the anatomical recurrence of the hernia. Definitions of recurrence include any evidence of the stomach above the diaphragm or more than 2 cm of herniation above the diaphragm.
  Endoscopic assessment: Esophagogastroduodenoscopy (EGD) is also used to identify recurrences.
  Recurrence rate= (number of recurrent patient/total arm patient) x100

CONTACTS AND LOCATIONS:
Locations (1):
- Asser Health Cluster, Abhā, 'Asir Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asti E, Lovece A, Bonavina L, Milito P, Sironi A, Bonitta G, Siboni S. Laparoscopic management of large hiatus hernia: five-year cohort study and comparison of mesh-augmented versus standard crura repair. Surg Endosc. 2016 Dec;30(12):5404-5409. doi: 10.1007/s00464-016-4897-7. Epub 2016 Apr 29. PMID 27129562
- [Background] Memon MA, Memon B, Yunus RM, Khan S. Suture Cruroplasty Versus Prosthetic Hiatal Herniorrhaphy for Large Hiatal Hernia: A Meta-analysis and Systematic Review of Randomized Controlled Trials. Ann Surg. 2016 Feb;263(2):258-66. doi: 10.1097/SLA.0000000000001267. PMID 26445468
- [Background] Zehetner J, Demeester SR, Ayazi S, Kilday P, Augustin F, Hagen JA, Lipham JC, Sohn HJ, Demeester TR. Laparoscopic versus open repair of paraesophageal hernia: the second decade. J Am Coll Surg. 2011 May;212(5):813-20. doi: 10.1016/j.jamcollsurg.2011.01.060. Epub 2011 Mar 23. PMID 21435915
- [Background] Morino M, Giaccone C, Pellegrino L, Rebecchi F. Laparoscopic management of giant hiatal hernia: factors influencing long-term outcome. Surg Endosc. 2006 Jul;20(7):1011-6. doi: 10.1007/s00464-005-0550-6. Epub 2006 Jun 8. PMID 16763927